CLINICAL TRIAL: NCT04563663
Title: Dose-response of Anteroposterior Mobilizations in Weight Bearing Talus Dorsiflexion in the Older Adult: Allegorized Clinical Trial
Brief Title: Dose-response of Anteroposterior Mobilizations in Weight Bearing Talus Dorsiflexion
Acronym: ANKLE_WBROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: KTV01
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Aging Problems
Keywords: Weight Bearing Dorsiflexion; Manual Therapy; Ankle; Dose-response

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- One session (Experimental): One session of talus posteriorization.
  Interventions: Procedure: Posteriorization of the talus.
- Two sessions (Experimental): Two sessions of talus posteriorization.
  Interventions: Procedure: Posteriorization of the talus.
- Three sessions (Experimental): Three sessions of talus posteriorization.
  Interventions: Procedure: Posteriorization of the talus.
- Four sessions (Experimental): Four sessions of talus posteriorization.
  Interventions: Procedure: Posteriorization of the talus.

INTERVENTIONS:
Procedure: Posteriorization of the talus. — Three sets of a 30-s grade IV anteroposterior mobilization.

SUMMARY:
Ankle mobility limitations are common in older adults. A possible treatment to restore joint mobility is manual therapy based on mobilization techniques, in this case, applied on the ankle joint. Previous research had proposed different treatment volumes (one to twelve sessions), but shown a different and non-consistent degree of effectiveness according to such factor. Therefore, this work aims to determine the dose-response relationship of manual therapy (talus mobilizations) on ankle range of motion in the older adult.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults.
* Limited ankle mobility (< 35 degrees).
* Over 60 years.

Exclusion Criteria:

* Not willing to participate or signing a consent form
* Lower limb injury in the three months prior to the study (ex. sprain)
* Diagnosed condition that may influence mobility assessments (i.e. stroke)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Treatment dose | Change from baseline to end of intervention (2 weeks) and follow-up (10 weeks)
  Number of sessions of experimental intervention needed to induce a clinically important gain in ankle mobility after the intervention. A baseline progression over 4.6º in the Lunge test will be considered clinically important (Powden, 2015), so that the number of sessions will be established when this threshold is exceeded (see secondary outcome) .

SECONDARY OUTCOMES:
The Lunge test | Change from baseline, to end of intervention (2 weeks) and follow-up (10 weeks)
  Weight bearing ankle dorsiflexion range of motion. This test will measure the maximum tilt of the tibia that a subject can perform while standing and bearing the weight on the limb without lifting the heel from the floor. A Baseline® Digital Inclinometer (Fabrication Enterprises Inc) will be used to assessed this outcome. Values below 35º indicate limited mobility. A baseline progression over 4.6º will be considered clinically important (Powden, 2015). This mobility gain will be used to determine the dose-response relationship: number of sessions of talus mobilizations needed to induce a clinically important gain in ankle mobility after the intervention (see primary outcome measure)

CONTACTS AND LOCATIONS:
Overall Officials: José-María Blasco, Study Director — University of Valencia; David Hernández-Guillén, Principal Investigator — University of Valencia; Catalina Tolsada-Velasco, Study Chair — University of Valencia
Locations (1):
- Universidad de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No